CLINICAL TRIAL: NCT04483570
Title: Urological Deterioration in Secondary Tethered Cord Syndrome and Clue to Detect It
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kwanjin Park, Associate Professor, Seoul National University Hospital
Other Study IDs: H-1809-029-969
Record Dates: First submitted 2020-07-07; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Neurogenic Bladder; Tethered Spinal Cord Syndrome
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Neural Tube Defects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Secondary Tethered Cord Syndrome: Children with signs of progressive deterioration in urological or neuroorthopedic system, and suspected Secondary Tethered Cord Syndrome (STCS) following primary untethering surgery.
  Interventions: Procedure: Redo-tethering operation

INTERVENTIONS:
Procedure: Redo-tethering operation

SUMMARY:
Secondary tethered cord syndrome (STCS) has been diagnosed with signs of progressive deterioration in urological or neuroorthopedic systems following primary tethering surgery. However, there is no convincing urological diagnostic clue for STCS.

DETAILED DESCRIPTION:
Tethered cord syndrome (TCS) refers to various problems involving neurologic, orthopedic, and urologic systems, seen as a result of chronic traction of the spinal cord in patients with spinal dysraphism. Evidence for neural injury is often assumed irreversible, so untethering is justified to maintain neural function and prevent further neural damage. Unfortunately, some patients experienced an aggravation of symptoms following untethering. The probable causes are assumed to be the neural injury before or during operation, which was revealed along with dysplastic neural function, neural compression by increasing syrinx and secondary tethered cord syndrome (STCS) in which postoperative neural adhesion or syrinx limit motion of spinal and elicit ischemic changes as the spine grows during puberty. The Secondary Tethered Cord Syndrome is reported as 19% of cases and causes significant progressive morbidities in those who affected.

Unfortunately, the detection of STCS is not as simple as it thought. Although magnetic resonance imaging (MRI) often reveals that the cord seems to get straightened, this does not necessarily mean that is a significant tethering or cord associated with progressive nerve damage. The variable course of progression and involvement of multiple systems such as lower extremity, bladder, bowel, and back would not allow a single specialist to draw conclusions about the presence of secondary tethered cord syndrome. Moreover, the untethering procedure of STCS may not always be safe and effective. Given the fact that a significant number of 'no improvement' or new onset complications following redo-untethering, the surgery could not be attempted without clear evidence. This explains the reason there is only a limited number of relevant studies so far.

In this study, it aims to delinate the genuine features of secondary tethered cord syndrome by selecting and analyzing only cases with symptom improvements. Furthermore, it described their natural history and time course of urological deterioration and characterized by the urodynamic changes before and after the redo-untethering.

ELIGIBILITY:
Inclusion Criteria:

- Children with signs of progressive deterioration in urological or neuroorthopedic system following primary untethering surgery.

Exclusion Criteria:

- Children without signs of progressive in urological or neuroorthopedic system following primary untethering surgery.

Ages: 3 Months to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with signs of progressive deterioration in urological or neuroorthopedic system, and suspected Secondary Tethered Cord Syndrome (STCS) following primary untethering surgery.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Pre-operative evaluation: Dysfunctional voiding | Baseline
  Evaluating any presence of urinary and fecal incontinence before the secondary tethered cord syndrome operation.
Pre-operative evaluation: Presence of Urinary Tract Infection (UTI) | Baseline
  Evaluating any presence of urinary and fecal incontinence before the secondary tethered cord syndrome operation
VUD (Video Urodynamic Studies) | Baseline
  Measuring maximal cystometric capacity, compliance, estimated bladder capacity before the operation of the secondary tethered cord syndrome.
VUD (Video Urodynamic Studies) | 1 year after the operation
  Measuring changes in maximal cystometric capacity, compliance, estimated bladder after the operation of the secondary tethered cord syndrome
VUD (Video Urodynamic Studies) | 2 years after the operation
  Measuring changes in maximal cystometric capacity, compliance, estimated bladder after the operation of the secondary tethered cord syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Kwanjin Park, MD, PHD, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No
Not plan to share IPD